CLINICAL TRIAL: NCT02888795
Title: Identification of Early Response to Hypertonic Dextrose Prolotherapy Markers in Knee Osteoarthritis Patients by an Inflammation-related Cytokine Array
Brief Title: Identification of Response to Hypertonic Dextrose Prolotherapy Markers in Knee Osteoarthritis Patients by Cytokine Array
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD2016-018
Record Dates: First submitted 2016-08-24; First posted 2016-09-05 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Osteoarthritis, Knee
Keywords: hypertonic dextrose prolotherapy; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hypertonic dextrose prolotherapy (Experimental)
  Interventions: Drug: hypertonic dextrose prolotherapy

INTERVENTIONS:
Drug: hypertonic dextrose prolotherapy — five intra-articular injection at 2-weeks intervals in weeks 0, 2, 4, 6, 8.

SUMMARY:
Hypertonic dextrose prolotherapy has been used in knee osteoarthritis (OA) clinically for a long time. However the study about the mechanism is scant. The question of biomarkers of knee OA cartilage response to hypertonic dextrose prolotherapy remains currently unresolved. On this basis, the aim of this study was to characterize the secreted protein factors behind the inflammatory potential involving the hypertonic dextrose prolotherapy of knee OA.

10~12 older than 65 years old knee OA patients will be recruited for clinical Western Ontario McMaster University Osteoarthritis (WOMAC) index, knee X ray evaluation and knee joint synovial fluid analysis before and after hypertonic dextrose prolotherapy. The expressions of inflammatory factors will be measured by a novel cytokine antibody array methodology. The study will evaluate inflammation-related cytokines in patients of knee joint synovial fluid. Human Cytokine Antibody Array that allows profiling synovial fluid production of anti and pro-inflammatory cytokines simultaneously. Altered levels of cytokine from the array membranes incubated with tissue lysates will quantitatively depict as a histogram for relative cytokine induction or reduction in the synovial fluid. The cytokines messenger ribonucleic acid levels will be quantified by quantitative reverse-transcription polymerase chain reaction and proteins expression was analyzed by Enzyme-Linked ImmunoSorbent Assay. The WOMAC Index, minimum joint space width, and Human Cytokine Antibody Array between before and after interventions will be compared. Differences between groups will be determined by the Mann-Whitney U test. For the synovial angiogenesis is accompanied with inflammatory feature in knee OA, associations between endothelial growth factor (VEGF) expression and VEGF isoforms pattern will be determined with the Spearman correlation.

ELIGIBILITY:
Inclusion Criteria:

* at least 6 months of symptomatic knee OA
* clinical criteria of moderate or moderate to severe knee OA ( the American Rheumatological Association grade II or III)

Exclusion Criteria:

* severe knee OA (grade IV)
* rheumatoid or other inflammatory arthritis
* received physiotherapy, oral NSAIDs, corticosteroids or anticoagulant, during previous 2 weeks prior the treatment
* received any knee intra-articular injections during previous one month prior the treatment
* poorly controlled diabetes mellitus with fasting blood sugar greater than 200 mg/dL-
* history of knee surgery
* dementia or psychological disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
Western Ontario McMaster University Osteoarthritis Index | change from baseline at week 10

SECONDARY OUTCOMES:
standing knee X ray posterior-anterior view | change from baseline at week 10
  the minimum joint space width (mJSW) of the medial and lateral compartment respectively of the tibio-femoral joint
protein array method for inflammatory factors | change from baseline at week 10
  Human Angiogenesis Antibody Array

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine & Rehabiliation, National Yang-Ming University Hospital, Yilan, Taiwan

IPD SHARING:
Plan to Share IPD: No
not all patients agreed to share primary data to person not related to study